CLINICAL TRIAL: NCT01011829
Title: A Randomized, Double-blind Trial of Varenicline Versus Placebo, in Conjunction With Cognitive Behavioral Therapy, for Methamphetamine Dependence
Brief Title: Varenicline vs Placebo for the Treatment of Methamphetamine Dependence
Acronym: RAVEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-18185-PII-3; P50DA018185 (NIH); DPMC (Other: NIH / NIDA)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-02

CONDITIONS: Methamphetamine Dependence; Substance Abuse; Methamphetamine Abuse
Keywords: methamphetamine; crystal meth; addiction; los angeles; medication; meth
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): Varenicline:
  0.5 mg daily for days 1-3
  0.5 mg twice daily for days 4-7
  1 mg twice daily from day 8 until end of week 8.
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): 8 weeks of daily matching oral placebo in tablet form
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline dosing will follow that which has been shown to be effective for cigarette smoking cessation. Varenicline dose will start at 0.5 mg daily for days 1-3, followed by 0.5 mg twice daily for days 4-7, followed by 1 mg twice daily from day 8 until completion of the medication period (end of week 8).
  Other Names: CHANTIX (tm)
  Arms: Varenicline
Drug: Placebo — Placebo dose will start at 0.5 mg (sugar pill) daily for days 1-3, followed by 0.5 mg twice daily for days 4-7, followed by 1 mg twice daily from day 8 until completion of the medication period (end of week 8).
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Methamphetamine (MA) abuse is the fastest growing drug problem in the United States and is responsible for significant public health complications, including HIV infection. As a result effective treatments for MA dependence are urgently needed. There are currently no efficacious medications for MA dependence, although results from preliminary randomized trials of bupropion for MA dependence found bupropion to be more effective than placebo, but only among subgroups of participants, including those with lower frequency of MA use at baseline. A growing body of preclinical and clinical studies suggest that cholinergic mechanisms play an important role in the neurobiology of MA and other stimulant dependence, such as nicotine dependence. Mechanistically, cholinergic medications may alleviate MA-associated cognitive dysfunction, thereby improving outcomes of treatment for MA dependence. Varenicline is a partial agonist at α4β2 nicotinic receptors and a full agonist at α7 nicotinic receptors that has been approved as an anti-cigarette smoking medication. In order to assess the potential efficacy of varenicline for methamphetamine dependence, we will perform a clinical trial to assess if varenicline compared to placebo results in greater:

1. reductions in methamphetamine use;
2. treatment retention;

DETAILED DESCRIPTION:
Methamphetamine (MA) abuse is the fastest growing drug problem in the United States and is responsible for significant public health complications, including HIV infection1. As a result effective treatments for MA dependence are urgently needed. There are currently no efficacious medications for MA dependence, although results from preliminary randomized trials of bupropion for MA dependence found bupropion to be more effective than placebo, but only among subgroups of participants, including those with lower frequency of MA use at baseline 2, 3. A growing body of preclinical and clinical studies suggest that cholinergic mechanisms play an important role in the neurobiology of MA and other stimulant dependence, such as nicotine dependence 4. Mechanistically, cholinergic medications may alleviate MA-associated cognitive dysfunction, thereby improving outcomes of treatment for MA dependence 5. Varenicline is a partial agonist at α4β2 nicotinic receptors and a full agonist at α7 nicotinic receptors that has been approved as an anti-cigarette smoking medication. In order to assess the potential efficacy of varenicline for methamphetamine dependence, we will perform a clinical trial to assess the following aims:

1. To determine if varenicline results in significantly greater reductions in methamphetamine use than placebo, as determined via the proportion of methamphetamine-free urine specimens provided by participants throughout treatment, when provided to methamphetamine dependent participants in conjunction with cognitive behavioral therapy.

   Exploratory Aim 1a. To determine whether reductions in methamphetamine use with varenicline versus placebo are greater among methamphetamine dependent participants with baseline light MA use (MA use on 18 or fewer of the past 30 days at baseline) versus heavy MA use (MA use on more than 18 of the past 30 days).

   Exploratory Aim 1b. To determine if varenicline results in a greater proportion of methamphetamine dependent participants achieving methamphetamine abstinence defined as self-reported MA abstinence, confirmed via urine drug screens (all available urine drug screens are MA-metabolite free and at least one urine drug screen available per week and no more than two missed visits between urine drug screens) during the final two weeks of the study medication period (weeks 7 and 8) relative to placebo when provided in conjunction with cognitive behavioral therapy.
2. To determine if varenicline results in significantly greater treatment retention than placebo among MA dependent participants when provided in conjunction with cognitive behavioral therapy.

To address these aims, we recruited 20 MA dependent participants who will be randomized to receive treatment with varenicline (n=10) or placebo (n=10) for 8 weeks, in combination with cognitive behavioral therapy, followed by 4 weeks of follow up observation.

Results of this study have the potential to provide additional safety data and to yield preliminary evidence that may support a fully powered late Phase II trial of the efficacy of varenicline for the treatment of methamphetamine dependence. Findings also have potential to provide insights into the influence of cognitive dysfunction, and medications with potential cognitive enhancing effects, on the pathogenesis of MA dependence and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. meet (Diagnostic and Statistical Manual of Mental Disorders) DSM-IV criteria for methamphetamine (MA) dependence;
3. seeking treatment for MA problems;
4. willing and able to comply with study procedures;
5. willing and able to provide written informed consent;
6. if female, not pregnant or lactating and willing to use an acceptable method of barrier birth control (e.g. condoms) during the trial.

Exclusion Criteria:

1. have a medical condition that, in the study physician's judgment, may interfere with safe study participation (e.g., active tuberculosis, unstable cardiac, renal, or liver disease, uncontrolled hypertension, unstable diabetes);
2. have a current neurological disorder (e.g., organic brain disease, dementia) or a medical history which would make study agent compliance difficult or which would compromise informed consent;
3. have a current major psychiatric disorder not due to substance abuse (e.g., schizophrenia, bipolar disorder) as assessed by the Structured Clinical Interview for DSM Disorders (SCID);
4. have a history of attempted suicide in the past 3 years and/or serious suicidal intention or plan in the past year as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS);
5. currently on prescription medication that is contraindicated for use with varenicline;
6. currently using any form of nicotine replacement therapy, due to potential interactions with varenicline;
7. have current dependence on cocaine, opiates, alcohol, or benzodiazepines as defined by DSM-IV;
8. have a history of alcohol dependence within the past three years;
9. have a history of sensitivity to varenicline or any other circumstances that, in the opinion of the investigators, would compromise participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoptaw, PhD, Principal Investigator — UCLA Dept of Family Medicine
Locations (1):
- UCLA Vine Street Clinic, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty treatment-seeking adults with current methamphetamine (MA) dependence were recruited through advertisements in newspapers, the internet, radio and community outreach from Nov 2009 to Feb 2010.
Pre-assignment Details: All potential subjects were consented and then completed study screening measures over a max. of six study visits in order to determine study eligibility. Subjects had to be over 18 years old, MA dependent, and looking for treatment with no Axis I disorder not related to substance abuse and have no contraindications for use of varenicline.
Groups:
- Varenicline: Varenicline dose will start at 0.5 mg daily for days 1-3, followed by 0.5 mg twice daily for days 4-7, followed by 1 mg twice daily from day 8 until completion of the medication period (end of week 8).
- Placebo (Sugar Pill): 8 weeks of daily matching oral placebo in tablet form
Period: Overall Study
Arm/Group | Varenicline | Placebo (Sugar Pill)
Started | 10 | 10
Completed | 6 | 1
Not Completed | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.4) | 35.1 (10.5) | 36.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in MA Positive Urine Drug Screens Among Participants Randomly Assigned to Receive Varenicline Versus Placebo.
Description: Urine samples, collected thrice weekly, were tested for metabolites of MA using radioimmunoassay. Each subject had a possible of 24 urine drug screens to provide during the 8 weeks of medication. An aggregate measure of urine drug screen results was calculated - the Treatment Effectiveness Score (TES) - which is the average of the sum of MA-free urine specimens provided during the treatment period by participants in each treatment condition.
Time Frame: 8-weeks
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: total MA-free urine drug screens
Units Other Than Participants: Urine drug screen results
Arm/Group | Varenicline | Placebo (Sugar Pill)
Number analyzed (Participants) | 10 | 10
Number analyzed (Urine drug screen results) | 24 | 24
total MA-free urine drug screens | 7.4 (10) | 2.3 (4.8)

2. Secondary Outcome: Retention (Completion)
Description: Retention was determined by the proportion of participants retained for the entire trial and time until drop-out.
Time Frame: 8-weeks
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo (Sugar Pill)
Number analyzed (Participants) | 10 | 10
participants | 6 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed at each study visit during the 8 weeks of treatment and in the follow up period (4 weeks).
Description: Subjects were questioned at each clinic visit about their general health. Any physical or clinical change or illness, whether or not considered study drug related, was recorded on the medical record chart and adverse event case report form. In case of an adverse event thought to reflect drug-related toxicity, evaluation and management ensued.
Arm/Group | Varenicline | Placebo (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=10) | Placebo (Sugar Pill) (N=10)
Insomnia (General disorders) | 3 (4) | 1 (1)
Irritability (Psychiatric disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Dysphoria (Psychiatric disorders) | 1 (1) | 1 (1)
Infection Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vivid Dreams (General disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression mental (Psychiatric disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Flushing (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Sex inhibition (General disorders) | 1 (1) | 0 (0)
Panic reaction (Psychiatric disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Immune system disorders) | 0 (0) | 1 (1)
Mental distress (Psychiatric disorders) | 2 (2) | 0 (0)
Urinary tract infection (General disorders) | 0 (0) | 1 (1)
Muscle ache (General disorders) | 0 (0) | 1 (1)
Paraesthesia (General disorders) | 0 (0) | 1 (1)
drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations in funding resulted in a small number of subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes